CLINICAL TRIAL: NCT06217900
Title: PROFOUND Study: Development and Validation of a Multi-cancer Early Detection Model Based on Peripheral Blood Multi-omic Analysis and Machine Learning: a Multicenter, Prospective, Observational, Case-control Study
Brief Title: a PROspective Case Control Study to Develop and Validate a Blood Test FOr mUlti-caNcers Early Detection（PROFOUND）
Acronym: PROFOUND
Status: Recruiting | Type: Observational
Sponsor: Shanghai Weihe Medical Laboratory Co., Ltd. (Industry)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROFOUND
Record Dates: First submitted 2023-12-28; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: cell-free DNA; methylation; cancer early detection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case arm: Participants with newly diagnosed cancer of lung, breast, digestive tract, urinary tract and etc.
- Control arm: Participants without a cancer diagnosis after routine cancer screening tests.

SUMMARY:
This study is a multi-center, case-control study aiming at developing and blinded testing machine learning-based multiple cancers early detection model by prospectively collecting blood samples from newly diagnosed cancer patients and individuals without confirmed cancer diagnosis.

DETAILED DESCRIPTION:
Blood samples from newly diagnosed cancer patients and individuals without confirmed cancer diagnosis will be prospectively collected to identify cancer-specific circulating signals through integrative multi-omic analysis. Based on the comprehensive molecular profiling, a machine learning-driven model will be trained and blinded validated independent through a two-stage approach in clinically annotated individuals. Approximately 10327 cancer patients will be enrolled in this study and early-stage cancer patients will be enriched to improve the model sensitivity on distinguishing cancers with favorable prognosis. Approximately 6339 age and sex matched controls will be included in model development, which are volunteers without a cancer diagnosis after routine cancer screening tests.

ELIGIBILITY:
Inclusion Criteria for Case Arm Participants:

* 40-74 years old
* Clinically and/or pathologically diagnosed cancer
* No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria for Case Arm Participants:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.5 °C) within 14 days prior to screen
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to screen
* Recipients of therapy in past 14 days prior to screen, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamide, hydrazine, arsenic trioxide
* Unsuitable for this trial determined by the researchers

Inclusion Criteria for Control Arm Participants:

* 40-74 years old
* Without confirmed cancer diagnosis
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria for Control Arm Participants:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.5 °C) within 14 days prior to screen
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to screen
* Recipients of therapy in the past 14 days prior to screen, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamide, hydrazine, arsenic trioxide
* Unsuitable for this trial determined by the researchers

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed cancers or individuals without confirmed cancer will be invited to participate in this case-control study by a designated consenting professional.
Sampling Method: Non-Probability Sample
Enrollment: 16666 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The performance of cfDNA methylation-based multiple cancers early detection model in case-control study | 12 months
  The sensitivity, specificity and tissue origin accuracy of cfDNA methylation-based multiple cancers early detection model in detecting cancer or non-cancer at 95% confidence interval.

SECONDARY OUTCOMES:
The performance of cfDNA methylation-based multiple cancers early detection model in early stage cancer cases | 12 months
  The sensitivity and tissue origin accuracy of cfDNA methylation-based multiple cancers early detection model in detecting stage I to II cancer at 95% confidence interval.
The performance of multi-omic-based multiple cancers early detection model in case-control study | 12 months
  The sensitivity, specificity and tissue origin accuracy of multi-omic-based multiple cancers early detection model in detecting cancer or non-cancer at 95% confidence interval.
The performance of different multi-cancer early detection models in different subgroups | 12 months
  The sensitivity and specificity of cfDNA methylation-based or multi-omic-based multiple cancers early detection model in different subgroups of the population (such as age, gender, cancer pathological classification, and clinical stage) at 95% confidence interval.

OTHER OUTCOMES:
To develop a questionnaire to evaluate the risk factors in the multi-cancer early screening | 12 months
  To develop a questionnaire to evaluate the high-risk factors in the multi-cancer early screening, including lung cancer, gastrointestinal cancer, gynecological cancer, urogenital neoplasms, etc.
To evaluate the performance of multi-omics early detection models in the population with suspected cancer | 12 months
  The sensitivity, specificity and tissue origin accuracy of multi-omic-based multiple cancers early detection model in in the population with suspected cancer at 95% confidence interval.
To simulate the positive predictive value and negative predictive value of different multi-cancer early detection models based on the cancer prevalence and staging data of individuals aged 40-75 years in China using multiple models | 12 months
  To simulate the positive predictive value and negative predictive value of different multi-cancer early detection models（cfDNA methylation-based or multi-omic-based)，based on the sensitivity, specificity and tissue origin accuracy，according to multi cancer prevalence and staging data of individuals aged 40-75 years in China.
To simulate the benefits of clinical utility and health economics using different multi-cancer early detection models | 12 months
  To simulate the stage-shift and incremental cost-effective ratio (ICER) benefit when compared to usual care (SOC screening) using Markov model based on MCED test performance
To explore biomarkers for cancer screening and construct a multimodal machine learning model based on multi-omics data | 12 months
  Exploring biomarkers in methylomics and fragmentomics，and constructing multimodal for multi-cancer early detection based on multiomics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, Principal Investigator — Peking University People's Hospital; Xiaohui Wu, Study Director — Shanghai Weihe Medical Laboratory Co., Ltd.
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No